CLINICAL TRIAL: NCT07032961
Title: Screening for Gastric Pathologies in Elderly and High-Risk Populations Using a Mobile Capsule Gastroscopy System: a Prospective, Multicenter, Population Based Cohort Study
Brief Title: A Cohort Study of Mobile Capsule Gastroscopy for Gastric Pathologies Screening
Status: Recruiting | Type: Observational
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Collaborators: Guangzhou First People's Hospital (Other); Second Affiliated Hospital of Guangzhou Medical University (Other); Guangdong Provincial Hospital of Traditional Chinese Medicine (Other)
Responsible Party: Sponsor
Other Study IDs: NFEC-2025-276
Record Dates: First submitted 2025-06-12; First posted 2025-06-24 (Actual); Last update posted 2025-07-04 (Actual); Status verified 2025-07

CONDITIONS: Gastritis; Gastric Dysplasia; Gastric Ulcer; Gastric Cancer; Gastric Mass
Keywords: Capsule Endoscopy; Prospective Study; screening
MeSH Terms: conditions — Gastritis; Stomach Ulcer; Stomach Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Enrolment Group: The enrolment group includes all subjects who will undergo MCG examination in the 'Gastric pathologies Screening Programme for the Elderly and High Risk Groups in Guangzhou Municipality'.
  Interventions: Other: Collect epidemiological, diagnostic, and follow-up data after MCG examination.

INTERVENTIONS:
Other: Collect epidemiological, diagnostic, and follow-up data after MCG examination. — MCG System: GICE-1000 Manufacturer: Guangzhou Side Medical Technology Co., Ltd.

SUMMARY:
The goal of this is to learn about the effectiveness and feasibility of a novel AI- assisted Mobile Capsule Gastroscopy (MCG) system for detecting gastric pathologies in elderly and high-risk populations.

The main question it aims to answer is:

Can MCG effectively detect gastric pathologies, including common gastric diseases, gastric cancer, and precancerous lesions, in elderly and high-risk individuals at community health centers?

Participants will:

Epidemiological, diagnostic, and post-MCG follow-up data generated during participants' involvement in the gastric pathologies public screening program will be collected.

DETAILED DESCRIPTION:
Gastric diseases-including atrophic gastritis, gastric polyps, peptic ulcers, submucosal lesions, gastric cancer, and precancerous conditions-have become a major global public health challenge. In China, the prevalence of gastric ulcers is as high as 17.2%, significantly higher than that in Western countries (4.1%) [1]. Gastric cancer also ranks among the top globally in both incidence and mortality, with approximately 400,000 new cases and over 300,000 deaths each year [2-3]. Notably, around 80% of patients are diagnosed at an advanced stage, and the 5-year survival rate is less than 30% [4]. Studies have shown that early gastric cancer, if detected and treated promptly, can achieve a 5-year survival rate of over 90% [5]. Moreover, if benign conditions such as atrophic gastritis and peptic ulcers are not treated in time, they may progress into precancerous lesions or even malignancies [6]. Therefore, early screening and accurate diagnosis are key to reducing the disease burden of gastric disorders.

Although esophagogastroduodenoscopy (EGD) is considered the gold standard for gastric disease screening [7-8], its invasive nature, associated patient discomfort, and reliance on skilled endoscopists and specialized equipment limit its accessibility. In China, the scarcity of endoscopic resources in primary care settings, combined with low patient compliance, further restricts screening coverage and increases the risk of missed diagnoses [9-10].

In recent years, capsule endoscopy has emerged as a valuable complementary tool for gastrointestinal disease screening due to its non-invasive and user-friendly nature [6,7]. Among its modalities, magnetically controlled capsule gastroscopy (MCCG) provides comprehensive gastric visualization, with reported sensitivity and specificity of 90% and 92%, respectively, for common gastric lesions. However, its reliance on expensive magnetic navigation systems and trained operators limits its widespread adoption in community-based screening programs [8].

To address these limitations, a novel mobile-controlled capsule gastroscopy (MCG) system being more accessible and not requiring costly external magnetic control was developed. It consists only of a disposable capsule and a wireless portable receiver. Participants can complete the examination independently in community health centers or at home by following video instructions via a smartphone app and adjusting their body positions to guide the capsule. An AI algorithm ensures complete gastric coverage in real time. The video can be viewed directly on the smartphone and transmitted to the cloud for remote diagnosis. The MCG system is non-invasive, user-friendly, and compatible with remote diagnosis, making it well suited for gastric disease screening in community health centers. Compared with MCCG, MCG enables fully autonomous operation without magnetic navigation, substantially reducing technical complexity and healthcare costs. However, its diagnostic accuracy and real-world feasibility in community-based populations have yet to be validated through prospective studies.

In 2025, the Guangzhou Municipal Health Commission issued the 'Gastric Pathologies Screening Programme for the Elderly and High Risk Groups in Guangzhou Municipality'. Organized by the Commission and led by Southern Medical University Nanfang Hospital, with participation from Guangzhou First People's Hospital, The Second Affiliated Hospital of Guangzhou Medical University, Guangdong Provincial Hospital of Traditional Chinese Medicine, and others, the program will conduct screening and surveillance of 10,000 elderly and high-risk individuals in community health centers across Guangzhou.

This prospective cohort study will collect epidemiological data, examination results, follow-up outcomes, and other relevant information from the screening program. The primary endpoint is the detection rate of gastric pathologies, including common conditions (such as atrophic gastritis, gastric ulcers, and submucosal tumors), gastric cancer, and precancerous lesions. The operational feasibility, safety, and acceptability of the MCG system in primary care settings will also be assessed. Findings are expected to provide scientific evidence to support the optimization of gastric disease prevention and control strategies at the municipal level.

1. Baseline Period

1. Record demographic data: gender, age
2. Record medical history and physical examination: including vital signs, anthropometric data (height and weight), comprehensive systemic assessment, history of smoking and alcohol use, Helicobacter pylori infection status, prior gastric pathologies, family history of gastric cancer, and mode of transportation to the clinic.

2. Diagnostic & Therapeutic Procedures

1. Record laboratory tests (if available), including complete blood count, stool analysis, prothrombin time, and the ¹³C/¹⁴C urea breath test.
2. Record the results of the MCG, the anatomical coverage of gastric regions, the rate of device failure and the overall image quality of the examination.
3. Record findings and therapeutic interventions from esophagogastroduodenoscopy (EGD) and histopathological biopsy results (if available).

3. Follow-up prognostic data

1. Record short-term follow-up data, including capsule endoscopy expulsion status, adverse events, referral outcomes, subsequent treatment, and patient compliance.
2. Record long-term follow-up data, including gastric pathologies incidence and survival rates of project participants.

3.1 Short-term follow-up will be conducted on Days 1, 3, and 14 following MCG.

1. Participants are instructed to inspect stool for capsule excretion and report the time of passage. If the capsule is not passed within 72 hours and gastrointestinal symptoms occur (e.g., constipation, abdominal pain), the research team will arrange clinical evaluation. Capsule retention will be conﬁrmed via abdominal X-ray or CT. Management may include prokinetic therapy or surgical retrieval as needed; the study will be discontinued post-retrieval in such cases.
2. All participants will receive a report summarizing the findings of the MCG examination. Researchers from community centers will follow up with individuals whose reports indicate significant gastric abnormalities to facilitate further medical management. Additionally, the overall study findings will be disseminated through publication in a peer-reviewed scientific journal.

3.2 Long-term follow-up will be conducted annually for a duration of five years through telephone interviews and/or routine monitoring at community health centers.

ELIGIBILITY:
Inclusion Criteria:

1.Provision of written informed consent; 2.Participants of the 'Gastric Pathologies Screening Programme for the Elderly and High Risk Groups in Guangzhou Municipality', the following are the criteria for inclusion in this public welfare programme:

1. Elderly cohort: Permanent residents of Guangzhou aged ≥60 years who have not undergone specialized gastric disease screening in the past three years;
2. Or high-risk cohort: Individuals aged ≥45 years who meet at least one of the following risk criteria:

   1. History of Helicobacter pylori infection (positive ¹³C/¹⁴C urea breath test);
   2. Prior diagnosis of chronic atrophic gastritis, gastric ulcer, neoplastic gastric polyps, hypertrophic gastritis, or pernicious anemia;
   3. Family history of gastric cancer (first-degree relative with a confirmed diagnosis);
   4. Long-term high-salt diet, smoking history (≥20 pack-years), or heavy alcohol consumption (100 mL of distilled spirits/day).

Exclusion Criteria:

1. Not considered by the investigator to be suitable for participation in this study.
2. Meets the exclusion criteria of the Public Welfare Programme. Individuals will be excluded if they meet any of the following conditions:

(1)Known allergy to medical polymer materials; (2)Psychiatric disorders that interfere with procedural cooperation; (3)Pregnancy or lactation; (4)Severe systemic comorbidities (e.g., cardiovascular, respiratory, neurological diseases) affecting examination tolerance; (5)Inflammatory bowel disease (Crohn's disease or ulcerative colitis) or gastrointestinal diverticulosis; (6)Known or suspected gastrointestinal malformations, obstructions, strictures, or fistulas; (7)Clinically significant dysphagia; (8)Acute abdominal symptoms (e.g., pain, vomiting, suspected bowel obstruction, or severe constipation); (9)History of major gastrointestinal surgery (e.g., esophagogastrostomy, gastrojejunostomy); (10)Physical debilitation precludes postural changes or concurrent severe illness; (11)Medically ineligible for abdominal procedures or refusal to undergo them; (12)Deemed unsuitable for MCG by the investigator; (13)Refusal to provide informed consent; (14)Any other condition judged by the investigator to make the individual unsuitable for study participation.

Min Age: 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 10,000 participants enrolled in the existing public welfare screening program: Gastric Pathologies Screening Programme for the Elderly and High Risk Groups in Guangzhou Municipality.
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2025-06-24 (Actual); Primary Completion 2026-10-31 (Estimated); Study Completion 2030-10-31 (Estimated)

PRIMARY OUTCOMES:
Detection Rate of Gastric Diseases Using Mobile Capsule Gastroscopy | At end of data collection phase (within 6 months of study launch)
  This measure assesses the proportion of participants in whom MCG identifies common gastric diseases, gastric cancer, or precancerous lesions.

SECONDARY OUTCOMES:
Safety of MCG | Within 14days after MCG procedure
  This outcome tracks the incidence and types of adverse events related to the MCG procedure, including capsule retention, discomfort, or complications requiring medical intervention.
Quality of MCG Examination | At end of data collection phase (within 6 months of study launch)
  The coverage rate of gastric anatomical regions, the device failure rate, image quality, and mucosal visibility will be evaluated for all MCG examinations.
  Coverage for each anatomical region and overall gastric coverage will be calculated as: Coverage rate = Number of Regions Adequately Visualized / Total Number of Anatomical Regions The calculation formula for the incidence of device failure is as follows: Device failure rate = Number of Cases with Device Failure / Number of Cases.
  A three-level grading scale (excellent / good / poor) will be used to objectively assess the following imaging quality indicators: clarity, field of view, image stability, structural and detail resolution, stereoscopic perception, overall image impression, intragastric cleanliness, gastric lumen distension, and mucosal visualization.
Procedural Compliance and Completion Rate | Immediately after MCG procedure
  This outcome evaluates the proportion of participants who successfully complete the MCG exam without technical failure or early termination.
Patient Satisfaction | Immediately after MCG procedure
  Participant-reported satisfaction with the MCG procedure, assessed via structured survey covering aspects such as comfort and convenience.
Cost-Effectiveness of MCG Screening | At end of data collection phase (within 6 months of study launch)
  Evaluates the cost per case of gastric pathologies detected using MCG versus conventional methods, using health economic metrics such as cost-effectiveness ratio and incremental cost-effectiveness ratio (ICER).
Diagnostic Agreement Between MCG and EGD (Kappa Value) | Within 30 days after MCG for participants referred for confirmatory EGD
  Measures the consistency of diagnosis between MCG and the gold-standard EGD in participants with suspicious MCG findings. The Kappa statistic will be calculated to quantify diagnostic agreement.

CONTACTS AND LOCATIONS:
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No